CLINICAL TRIAL: NCT02980471
Title: Comparison of Compensatory Reserve Index to Changes in Stroke Volume and Intravascular Volume
Status: Completed | Type: Observational
Sponsor: Flashback Technologies (Industry)
Collaborators: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00049209
Record Dates: First submitted 2016-11-30; First posted 2016-12-02 (Estimated); Last update posted 2016-12-02 (Estimated); Status verified 2016-12

CONDITIONS: Hemorrhage
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Pulse Oximeter — Blood removal and reintroduction as measured by the plethysmograph of a pulse oximeter

SUMMARY:
The purpose of this study is to demonstrate the correlation of the Compensatory Reserve Index (CRI) numeric and graphical trend readings to intravascular volume changes as compared to graded blood loss (removal of 20% of estimated total blood volume in ~333 mL aliquots) and to stroke volume as measured by the Nexfin monitor during the same graded blood removal period. Enrollment includes both men and women.

DETAILED DESCRIPTION:
Sequential Blood Loss: Blood loss will be simulated by withdrawal of 20% of estimated total blood volume. Estimated total blood volume for men = 75 mL/kg and for women = 65 mL/kg. The calculated target withdrawal volume is also consistent with an allowable estimated blood loss equation assuming a starting hematocrit (hct) of approximately 45% in males and 40% in females, where the expected drop in hct for this volume withdrawn is 7 percentage points in males and 6 percentage points in females. An actual drop in hct may not be observed in this study due to the relatively expedient removal of blood and no simultaneous administration of fluids (i.e., no "hemodilution" with crystalloid). Blood will be removed in aliquots up to ~333 mL. For safety, men will have no more than 4 units of blood removed (1,333 mL) and women will have no more than 3 units of blood removed (1,000 mL).

The blood will be withdrawn via the venous catheter and we anticipate that it will take 15-20 min for each stage of blood withdrawal to occur. A total of 3 aliquots will be withdrawn over approximately sixty minutes in women and 4 aliquots withdrawn over 80 minutes in men. The blood will be stored using preservatives and anticoagulation procedures similar to those used for perioperative hemodilution and/or intraoperative cell saver. The blood will remain in the study room until it is re-infused. We will use standard "auto-transfusion" blood collection equipment identical to that used in the ORs for perioperative hemodilution techniques. The blood will be drained by gravity from an indwelling vascular catheter into anti-coagulant preservative solution using tubing and bags systems provided by the autologous transfusion team that we routinely work with in the ORs. For the first several studies we will schedule them at a time when auto-transfusion OR personnel can be present and after that the anesthesiologists will be directly involved in drawing the blood, subsequent handling and reinfusion. The blood will never leave the autologous transfusion bag and a closed system will be used. The blood will be held at room temp with gentle agitation for ~60-80 minutes and then re-infused over 60-80 minutes via a large bore IV; monitoring will continue during reinfusion. Following completion of the reinfusion subjects will de-instrumented and observed in the physiology lab for two hours.

ELIGIBILITY:
Inclusion Criteria:

* • Ages 18-55.

  * Physical status: Healthy ASA Class 1.
  * Male or female.
  * Screening hemoglobin > 13.5 g/dl and hematocrit > 39% for males
  * Screening hemoglobin > 12 g/dl and hematocrit > 35% for females
  * BMI <30
  * Ability to provide written informed consent.
  * Willing and able to comply with study procedures

Exclusion Criteria:

* • Subjects with injuries, deformities or abnormalities that may prevent proper application of the device under test

  * Subjects with known respiratory conditions (uncontrolled asthma, head cold, flu, pneumonia / bronchitis, respiratory distress / respiratory or lung surgery, emphysema, COPD, lung disease),
  * Subjects with history of cardiovascular disease, hypertension, diabetes or any other diseases/conditions that might negatively influence their ability to tolerate moderate but temporary blood loss.
  * Obese subjects (BMI>30)
  * Smoker.
  * Subjects on drugs of any type (except oral contraceptives).
  * Female subjects that are actively trying to get pregnant or are pregnant.
  * Subjects taking blood thinners or medications with antiplatelet factors.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Twenty healthy volunteers between the ages of 18 and 55, men and women, American Society of Anesthesiology "class 1" health status.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2014-03; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Comparison of CipherOx trend to blood removal for trending intravascular volume | 1 hour
  comparison of CipherOx reading trend before removal of blood, post 330mL, 660mL and 1,000mL blood removal for trending intravascular volume change

IPD SHARING:
Plan to Share IPD: No